CLINICAL TRIAL: NCT00641693
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel Group, Phase II Study to Assess the Efficacy and Safety of RHINOCORT AQUA (Budesonide) Nasal Spray 16mg, 32mg and 64mg Per Day Versus Placebo in Paediatric Subjects Ages 2-5 Years Old With Allergic Rhinitis.
Brief Title: Assess the Efficacy and Safety of Rhinocort Aqua
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5360C00703; SD-005-0703
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis; Paediatric; Nasal symptoms; Congestion; Rhinorrhea; Sneeze; budesonide; Rhinocort AQUA
MeSH Terms: conditions — Rhinitis, Allergic; Rhinorrhea; Sneezing | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Nasal Spray
  Interventions: Drug: Budesonide
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide — 16mg Nasal Spray
  Other Names: Rhinocort AQUA
  Arms: 1
Drug: Budesonide — 32mg Nasal Spray
  Other Names: Rhinocort AQUA
  Arms: 1
Drug: Budesonide — 64mg Nasal Spray
  Other Names: Rhinocort AQUA
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to compare Rhinocort with placebo in pediatric subjects aged 2-5 years with allergic rhinitis to study effects on nasal symptoms such as sneezing, runny and stuffy noses.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator, is a candidate for treatment with nasal steroids based on a history of either a) inadequate control of symptoms with antihistamines, decongestants and/or immunotherapy, or b) prior successful treatment with nasal steroids.
* A documented history of allergic rhinitis and a positive response to a skin prick test at Visit 1 or within the last 12 months for allergens that must be present in the subject's environment for the duration of the study.
* At randomisation having nasal symptom scores as defined by the protocol.

Exclusion Criteria:

* Primary or secondary adrenal insufficiency
* Nasal candidiasis, rhinitis medicamentosa, acute or chronic sinusitis, influenza, upper respiratory tract infection or structural abnormalities of the nose (e.g., septal deviation, nasal polyps) symptomatic enough to cause significant nasal obstruction as judged by the investigator.
* A diagnosis of asthma requiring treatment as specifies in the protocol.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 650 (Estimated)
Dates: Start 2004-04; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
To compare Rhinocort with placebo to compare effects on nasal symptoms such as sneezing, runny and stuffy noses as assessed by caregivers. | At 2 weeks

SECONDARY OUTCOMES:
Safety assessment via adverse events and clinical measurements | At 1 & 2 weeks
To assess efficacy of Rhinocort via the physician and caregivers assessments | At 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Liza O'Dowd, MD, Study Director — AstraZeneca; Bertil Andersson, Study Director — AstraZeneca